CLINICAL TRIAL: NCT04499222
Title: Assessment of Tube Position According to the Changes of Neck Position Between Two Different Types of Nasotracheal Tubes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2020-0654
Record Dates: First submitted 2020-07-30; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Nasotracheal Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Portex (Experimental): usage of PORTEX POLAR [Smiths Medical International, Hythe, United Kingdom] nasotracheal tube
  Interventions: Device: Portex
- Mallinckrodt (Active Comparator): usage of Mallinckrodt TaperGuard [Covidien, Ireland] nasotracheal tube
  Interventions: Device: Mallinckrodt

INTERVENTIONS:
Device: Portex — nasotracheal intubation with PORTEX POLAR [Smiths Medical International, Hythe, United Kingdom] nasotracheal tube.
  Arms: Portex
Device: Mallinckrodt — nasotracheal intubation with Mallinckrodt TaperGuard [Covidien, Ireland] nasotracheal tube.
  Arms: Mallinckrodt

SUMMARY:
The aim of this study is to evaluate the appropriateness of the two kinds of nasotracheal tube (PORTEX POLAR [Smiths Medical International, Hythe, United Kingdom], Mallinckrodt TaperGuard [Covidien, Ireland]) depth in neutral, extended and flexed neck position when the upper border of the cuff of endotracheal tube is located 3cm below the vocal cords in neutral neck position.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients who undergoes elective surgery under general anesthesia with nasotracheal intubation

Exclusion Criteria:

1. Patients under 20 years old
2. Patients with ASA class IV or higher
3. Pregnant women
4. Patients receiving emergency surgery
5. Patients who have nasal disease or who undergo nose surgery because of nasal disease
6. Patient with craniofacial anomaly
7. Patients with impaired cervical motion
8. Patients who can not read the consent form or are not fluent in Korean (illiterate, foreigner)
9. Patients who refused the clinical trial Patients with dementia or cognitive impairment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The adequacy of nasotracheal tube tip location in neutral, extended and flexed neck position | 1 minute after nasotracheal intubation
  1. whether the tube tip is located above the carina in neutral, extended and flexed neck position when the upper border of the cuff of endotracheal tube is fixed 3cm below the vocal cords (in neutral neck position).
  2. the distance from the carina to the tube tip in neutral, extended and flexed neck position when the upper border of the cuff of endotracheal tube is fixed 3cm below the vocal cords (in neutral neck position).

SECONDARY OUTCOMES:
The adequacy of nasotracheal tube cuff location in extended and flexed neck position | 1 minute after nasotracheal intubation
  whether the tube cuff is located below the vocal cords in extended and flexed neck position when the upper border of the cuff of endotracheal tube is fixed 3cm below the vocal cords in neutral neck position.
The adequacy of nasotracheal tube length | 1 minute after nasotracheal intubation
  whether the tube cuff cannot be located 3cm below the vocal cords owing to short length of nasotracheal tube.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No